CLINICAL TRIAL: NCT00094861
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Palifermin (Recombinant Human Keratinocyte Growth Factor) in the Reduction of Dysphagia in Patients Receiving Concurrent Chemoradiotherapy Followed by Consolidation Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study to Evaluate Palifermin in the Reduction of Dysphagia in Patients With Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030185
Record Dates: First submitted 2004-10-27; First posted 2004-10-27 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Dysphagia; Non-Small Cell Lung Cancer; Lung Cancer
Keywords: dysphagia; palifermin, KGF; chemoradiotherapy; NSCLC, non-small cell lung cancer; lung cancer; supportive care; clinical trial; consolidation chemotherapy; radiotherapy
MeSH Terms: conditions — Deglutition Disorders; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Fibroblast Growth Factor 7; Radiotherapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single intravenous (IV) dose of placebo administered 3 days before the initiation of concurrent chemo/radiotherapy, then once weekly during Weeks 1 through 6, typically for a total of 7 doses. Concurrent radio/chemotherapy was given as follows:
  * standard radiotherapy 2 Gy once daily x 30 to 33 fractions (6 to 7 weeks) for a total target dose of 60 to 66 Gy
  * paclitaxel 50 mg/m^2 intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy)
  * carboplatin dosed at an area under the curve (AUC) 2.0 IV on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy).
  Participants subsequently received two 21-day cycles of consolidation chemotherapy with paclitaxel 225 mg/m^2 and carboplatin dosed at AUC 6.0.
  Interventions: Drug: Placebo; Radiation: Radiotherapy; Drug: Paclitaxel; Drug: Carboplatin
- Palifermin (Experimental): Participants received a single IV dose of palifermin at 180 μg/kg administered 3 days before the initiation of concurrent chemo/radiotherapy, then once weekly during Weeks 1 through 6, typically for a total of 7 doses. Concurrent radio/chemotherapy (administered for 6 to 7 weeks) was given as follows:
  * standard radiotherapy 2 Gy once daily x 30 to 33 fractions (6 to 7 weeks) for a total target dose of 60 to 66 Gy
  * paclitaxel 50 mg/m^2 IV infusion on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy)
  * carboplatin dosed at an area under the curve (AUC) 2.0 IV on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy).
  Participants subsequently received two 21-day cycles of consolidation chemotherapy with paclitaxel 225 mg/m^2 and carboplatin dosed at AUC 6.0.
  Interventions: Drug: Palifermin; Radiation: Radiotherapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Palifermin
  Other Names: Recombinant Human Keratinocyte Growth Factor; rHuKGF; Kepivance
  Arms: Palifermin
Drug: Placebo
  Arms: Placebo
Radiation: Radiotherapy
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The purpose of this study is to determine if palifermin will reduce the incidence of dysphagia in patients receiving concurrent chemoradiotherapy followed by consolidation chemotherapy for treatment of unresectable stage III Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
During the acute dysphagia evaluation phase (the period lasting from the administration of the first dose of investigational product through Week 12 (or up to Week 16 if dysphagia is not resolved to CTCAE v3.0 grade ≤ 1 by Week 12) participants underwent acute dysphagia assessments twice weekly. All participants were followed for disease progression, second primary tumors, other malignancies, and overall survival until death or loss to follow-up during the long term follow-up (still ongoing).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically proven diagnosis of NSCLC
* Unresectable (locally advanced) stage IIIa or IIIb disease
* Initial radiotherapy field of treatment to encompass greater than or equal to 30% of the esophagus
* Life expectancy greater than or equal to 6 months
* Estimated weight loss less than or equal to 10% in the 3 months before study randomization
* Measurable disease
* 18 years of age or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Hemoglobin (hgb) greater than or equal to 10 g/dL without transfusional support or growth factor use in the 4 weeks before study randomization
* Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L without growth factor use in the 2 weeks before study randomization
* Platelet count greater than or equal to 100 x 10^9/L
* Serum bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN)
* Serum creatinine less than or equal to 2.0 mg/dL (Note: Patients with a serum creatinine greater than or equal to 1.4 and less than or equal to 2.0 mg/dL must demonstrate a 24-hour urinary creatinine clearance greater than or equal to 50 mL/min)
* Females of childbearing potential: negative serum or urine pregnancy test
* Patient must give written informed consent before participating in any study-specific procedure, randomization, or receiving investigational product.
* Patients with reproductive capability must agree to practice adequate contraception methods.

Exclusion Criteria:

* Metastatic disease (M1)/stage 4 NSCLC
* Pleural or pericardial effusion greater than 100 ml in volume as documented by appropriate imaging (positron emission tomography [PET], computed tomography [CT] scan or ultrasound). If an effusion greater than 100 ml is documented by cytology to be free from malignancy and the investigator feels the patient is capable of receiving chemo/radiotherapy for their primary disease/ NSCLC, the investigator should discuss the patient with the study physician at Amgen. Effusions smaller than 100 ml would be acceptable, unless the investigator suspects that the effusion is malignant, in which case the effusions should be evaluated by cytology. Sponsor approval must be obtained before patient is randomized.
* Plan to remove the tumor surgically before completing the protocol chemo/radiotherapy course
* Shielding of any part of the esophagus during radiotherapy (including posterior spinal cord shielding)
* Prior chemotherapy, radiotherapy, or surgery for NSCLC
* Prior invasive malignancy during the past 3 years other than non-melanomatous skin cancer. Note: Patients with prior surgically-cured malignancies [eg, stage I breast cancer or prostate cancer, in-situ carcinoma of the cervix, etc] are not excluded; however, sponsor approval must be obtained before patient is randomized.
* Presence or history of dysphagia or conditions predisposing to dysphagia (eg, uncontrolled gastroesophageal reflux disease [GERD], dyspepsia, etc)
* History of pancreatitis
* Four weeks or less since completion of treatment using an investigational product/device in another clinical study or presence of any unresolved toxicity from previous treatment
* Previous treatment on this study or with a fibroblast growth factor
* Known to be sero-positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV)
* Pregnant or breastfeeding women
* Known sensitivity to E. coli derived products
* Compromised ability of the patient to give written informed consent and/or to comply with study procedures
* Refusal to sign an informed consent form to participate in this study, and sign the hospital information release form, if applicable
* Unwilling or unable to complete the patient reported outcome (PRO) questionnaires
* Psychological, social, familial, or geographical reasons that would prevent regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 06 January 2005 until 20 December 2007 (last participant's last visit for the acute dysphagia evaluation phase). At the time of this report, the long-term safety follow-up period is ongoing.
Pre-assignment Details: 100 patients were initially enrolled at 25 sites, however, data from one site could not be used and is excluded from this results analysis.
Groups:
- Placebo: Participants received a single intravenous (IV) dose of placebo administered 3 days before the initiation of concurrent chemo/radiotherapy, then once weekly during Weeks 1 through 6, for a total of 7 doses. Concurrent radio/chemotherapy was given as follows:
  * standard radiotherapy 2 Gy once daily x 30 to 33 fractions (6 to 7 weeks) for a total target dose of 60 to 66 Gy
  * paclitaxel 50 mg/m^2 intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy)
  * carboplatin dosed at an area under the curve (AUC) 2.0 IV on Days 1, 8, 15, 22, 29, 36 (and day 43 for those receiving 66 Gy).
  Participants subsequently received two 21-day cycles of consolidation chemotherapy with paclitaxel 225 mg/m^2 and carboplatin dosed at AUC 6.0.
Period: Overall Study
Arm/Group | Placebo | Palifermin
Started | 46 | 49
Participants Treated | 46 | 48
Completed | 28 (Participants who completed the acute dysphagia evaluation phase) | 40 (Participants who completed the acute dysphagia evaluation phase)
Not Completed | 18 | 9
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 4 | 2
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received a single intravenous (IV) dose of placebo administered 3 days before the initiation of concurrent chemo/radiotherapy, then once weekly during Weeks 1 through 6, typically for a total of 7 doses.
- Palifermin: Participants received a single IV dose of palifermin at 180 μg/kg administered 3 days before the initiation of concurrent chemo/radiotherapy, then once weekly during Weeks 1 through 6, typically for a total of 7 doses.
- Total: Total of all reporting groups
Arm/Group | Placebo | Palifermin | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.7) | 61.6 (9.8) | 62.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 32 | 34 | 66
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Causcasian | 43 | 43 | 86
  Black or African-American | 2 | 2 | 4
  Hispanic or Latino | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Japanese | 0 | 1 | 1
  Other | 0 | 1 | 1
Disease Stage [Number; unit: participants] — American Joint Committee on Cancer (AJCC) disease stage.
  participants
    Stage 3A | 14 | 19 | 33
    Stage 3B | 32 | 30 | 62
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; Grade 5: Dead.
  participants
    Grade 0 | 21 | 21 | 42
    Grade 1 | 23 | 26 | 49
    Grade 2 | 2 | 2 | 4
Weight Loss Over Last 3 Months [Number; unit: participants]
  < 5% | 35 | 37 | 72
  5 - 10% | 11 | 12 | 23
Randomization Strata [Number; unit: participants] — Baseline disease stage (3A or 3B), Baseline ECOG performance status (0-1 or 2), Estimated weight loss in 3 months before study (<5% or 5-10%)
  participants
    3A, 0-1, <5% | 10 | 11 | 21
    3A, 0-1, 5-10% | 4 | 6 | 10
    3A, 2, <5% | 1 | 2 | 3
    3A, 2, 5-10% | 1 | 0 | 1
    3B, 0-1, <5% | 24 | 25 | 49
    3B, 0-1, 5-10% | 6 | 5 | 11
    3B, 2, <5% | 0 | 0 | 0
    3B, 2, 5-10% | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Dysphagia
Description: Participants underwent acute dysphagia assessments twice weekly during Weeks 1 through 7, and twice weekly thereafter (Weeks 8 through 12) and once weekly after Week 12 until dysphagia resolved to grade ≤ 1 but not beyond Week 16. Dysphagia (difficulty swallowing) was graded using the Common Terminology Criteria for Adverse Events, Version 3.0 (CTCAE v3.0) dysphagia scale according to the following:
  Grade 1: Symptomatic, able to eat regular diet; Grade 2: Symptomatic and altered eating/swallowing (e.g., altered dietary habits, oral supplements), IV fluids indicated <24 hours; Grade 3: Symptomatic and severely altered eating/swallowing (e.g., inadequate oral caloric or fluid intake), IV fluids, tube feedings, or total parenteral nutrition (TPN) indicated ≥24 hours; Grade 4: Life-threatening consequences (e.g., obstruction, perforation).
Time Frame: Start of treatment through Week 16
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 46 | 49
participants
  Yes | 32 | 30
  No | 13 | 18
  No assessment | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.3550, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants with no assessments were assumed as having grade ≥ 2 dysphagia in hypothesis testing; Stratified by disease stage, ECOG performance status, and estimated weight loss in the 3 months before study randomization; Chi-Square Statistic = 0.8553

2. Secondary Outcome: Duration of Grade 2 or Higher Dysphagia
Description: Duration of grade 2 or higher dysphagia was calculated in days from the onset (first occurrence of grade ≥ 2) to the resolution (grade ≤ 1 after the last grade ≥ 2) of dysphagia.
  Participants with no assessments were assumed as having grade ≥ 2 dysphagia and with a duration of the mean duration of all participants.
Time Frame: Start of treatment through Week 16
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 46 | 49
days | 32.4 (30.1) | 25.3 (28.0)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.3189, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for mean score difference using modified ridit score; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.9936

3. Secondary Outcome: Maximal Dysphagia Grade
Description: The mean maximal grade of dysphagia for each participant during the study. Dysphagia (difficulty swallowing) was graded using the Common Terminology Criteria for Adverse Events, Version 3.0 (CTCAE v3.0) dysphagia scale according to the following:
  Grade 1: Symptomatic, able to eat regular diet; Grade 2: Symptomatic and altered eating/swallowing (e.g., altered dietary habits, oral supplements), IV fluids indicated <24 hours; Grade 3: Symptomatic and severely altered eating/swallowing (e.g., inadequate oral caloric or fluid intake), IV fluids, tube feedings, or total parenteral nutrition (TPN) indicated ≥24 hours; Grade 4: Life-threatening consequences (e.g., obstruction, perforation).
Time Frame: Start of treatment through Week 16
Population: Full analysis set participants with dysphagia assessments.
Measure: Mean (Standard Deviation); unit: grade
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 45 | 48
grade | 1.9 (1.0) | 1.8 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.5086, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants with no assessments were assumed as having grade 5 dysphagia in hypothesis testing; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.4370

4. Secondary Outcome: Number of Participants With Severe (Grade 3 or Higher) Dysphagia
Description: as for outcome 1
Time Frame: Start of treatment through Week 16
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 46 | 49
participants
  Yes | 13 | 11
  No | 32 | 37
  No assessment | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.4976, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants with no assessments were assumed as having grade ≥ 3 dysphagia in hypothesis testing; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.4600

5. Secondary Outcome: Number of Participants With Unplanned Breaks in Radiotherapy
Description: The number of participants with unplanned breaks in radiotherapy of ≥ 5 days or who discontinued radiotherapy during Week 1 to Week 6.
Time Frame: Week 1 to Week 6
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 46 | 49
participants
  Yes | 15 | 9
  No | 29 | 38
  Did not receive radiotherapy | 2 | 2
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.1115, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association. Participants who never received radiotherapy were assumed to have unplanned breaks; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = -2.5325

6. Secondary Outcome: Maximal Eastern Cooperative Oncology Group (ECOG) Performance Status Increase
Description: Maximal increase from Baseline in Eastern Cooperative Oncology Group (ECOG) performance status. ECOG is a scale to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; Grade 5: Dead.
Time Frame: Baseline through Week 12
Population: Full analysis set participants with available ECOG data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 44 | 46
units on a scale | 1.5 (1.3) | 0.9 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.0621, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel (CMH) test for mean score difference using modified ridit score. Participants without any ECOG assessment post baseline were assumed to have ECOG status of 5 in the CMH test; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 3.4812

7. Secondary Outcome: Number of Participants Hospitalized
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 46 | 49
participants
  Hospitalized | 31 | 34
  Not hospitalized | 15 | 15
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = 0.8639, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for general association; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 0.0294

8. Secondary Outcome: Maximal Body Weight Loss
Description: Maximal weight loss observed from Baseline through to Week 12.
Time Frame: Baseline through Week 12
Population: Full analysis set with available data
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Palifermin
Number analyzed (Participants) | 42 | 45
kilograms | 4.63 (4.13) | 5.44 (4.33)
Statistical Analysis 1: Comparison: Placebo vs Palifermin; Test type: Superiority or Other; p = 0.1996, Cochran-Mantel-Haenszel — Generalized Cochran-Mantel-Haenszel test for mean score difference using modified ridit score; [statistical method as in outcome 1, analysis 1]; Chi-Square Statistic = 3.1414

ADVERSE EVENTS:
Time Frame: From baseline up to Week 12
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Palifermin
Serious Adverse Events (participants affected / at risk) | 30/46 | 21/48
Other Adverse Events (participants affected / at risk) | 45/46 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Palifermin (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 7
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Vision blurred (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 4
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Chest discomfort (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 2 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | Palifermin (N=48)
Anaemia (Blood and lymphatic system disorders) | 21 | 27
Leukopenia (Blood and lymphatic system disorders) | 8 | 18
Neutropenia (Blood and lymphatic system disorders) | 11 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 10
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 9 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 23 | 25
Oesophagitis (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 11 | 10
Asthenia (General disorders) | 5 | 9
Chest pain (General disorders) | 4 | 7
Fatigue (General disorders) | 14 | 19
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 4 | 2
Pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 9 | 8
Pneumonia (Infections and infestations) | 1 | 5
Radiation skin injury (Injury, poisoning and procedural complications) | 6 | 10
Weight decreased (Investigations) | 7 | 6
Anorexia (Metabolism and nutrition disorders) | 8 | 13
Dehydration (Metabolism and nutrition disorders) | 6 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 5 | 6
Dysgeusia (Nervous system disorders) | 3 | 8
Headache (Nervous system disorders) | 3 | 4
Hypoaesthesia (Nervous system disorders) | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 4
Paraesthesia (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 4
Anxiety (Psychiatric disorders) | 6 | 3
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 10
Erythema (Skin and subcutaneous tissue disorders) | 2 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Flushing (Vascular disorders) | 0 | 5
Thrombophlebitis (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits sponsor a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Sponsor may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, investigator agrees not to publish any results before the first multi-center publication.